CLINICAL TRIAL: NCT05767944
Title: Wide-Awake Local Anesthesia No Tourniquet (WALANT) Versus Regional Anesthesia With Tourniquet for Hand Flexor Tendon Repair Surgeries in Adults
Brief Title: Awake Local Anesthesia Infiltration Compared to Regional Nerve Block for Hand Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS 242/2022
Record Dates: First submitted 2023-01-26; First posted 2023-03-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: Anaesthesia Conduction
Keywords: WALANT (Wide-Awake Local Anesthesia No Tourniquet ); Regional Anesthesia; Hand flexor Tendon Repair; Supra-clavicular brachial plexus block; Hand surgery
MeSH Terms: interventions — Brachial Plexus Block

STUDY DESIGN:
Intervention Model Description: patients were allocated to one of two groups. one received WALANT (with no tourniqut) & the other (control) group received supra-clavicular block (with tourniquet). Groups were compared for anaesthesia efficiency
Who Masked: Outcomes Assessor
Masking Description: For those assessing & providing postoperative analgesia (secondary outcome)they are blind to the used anaesthetic technique .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wide Awake Local Anesthesia (WALANT) (Experimental): Study arm: (WALANT) patient received local anaesthesia (25ml of 2%lidocaine with 0.5 ml of adrenaline (1mg/mL) and 5 ml of 8.4% of sodium bicarbonate. the final 50 ml mixture contained 10 mg/ml Lidocaine and adrenaline 1:100,000 concentration) infiltration along rays at site of surgery (15 ml or more per ray (150 mg lidocaine) by 27G needle, 10 ml (or more) in the palm, then 2 ml in the proximal and middle phalanges and 1 ml in the distal phalanx (if required )) for hand flexor tendons repair.
  Interventions: Other: local anaesthesia infiltration
- Supra Clavicular- Brachial Plexus Block (SC-BPB) (Active Comparator): Control arm:(SC-BPB): ultrasound-guided injection of local aesthetics (15 mL of 2% lidocaine and 15 mL of 0.5% bupivacaine were injected incrementally over 3-5 min) at supra-clavicular level where brachial plexus trunks are located this will provide anesthesia for the whole upper limb distal to shoulder joint.
  Interventions: Other: brachial plexus block

INTERVENTIONS:
Other: local anaesthesia infiltration — Infiltration of 150 mg of lidocaine solution per ray at site of surgical incision for flexor tendon repair in the palm, the 2 proximal & distal phalanges
  Arms: Wide Awake Local Anesthesia (WALANT)
Other: brachial plexus block — ultrasound-guided infiltration of local aesthetics around brachial plexus trunks & divisions
  Arms: Supra Clavicular- Brachial Plexus Block (SC-BPB)

SUMMARY:
The study trying to fined out the best anaesthesia technique for hand flexor procedures which provide efficient anaesthesia while providing adequate surgical field exposure & less blood loss

DETAILED DESCRIPTION:
The current study compared patients scheduled for hand surgical procedures using wide awake local anaesthetic infiltration to those receiving supra-clavicular brachial plexus block. the comparison including adequacy of pain control, blood loss, patient satisfaction, time & skills needed to provide aesthetic technique.

ELIGIBILITY:
Inclusion Criteria:

* Participants were included if they were to be scheduled for Flexor tendon repair (Interventions involving flexor tendons of the wrist (Flexor Carpi Ulnaris (FCU), Flexor Carpi Radialis (FCR), and/or Palmaris Longus PL), fingers (flexor digitorum Profundus FDP and/or Flexor Digitorum Superficialis FDS) and thumb (Flexor Pollicis Longus FPL)), aged 18 years or over & of ASA physical status I or II.

Exclusion Criteria:

* Participants were excluded if they were (American society of Anaesthesia) ASA physical status III or IV, refusal of anaesthetic procedure or refuse to participation in the study, documented hypersensitivity to lidocaine, compromised peripheral circulation (Patients with previous vascular injury, vasculitis, Buerger's disease, and scleroderma), evidence of infection at injection site, patients with ischemic heart disease or psychiatric illness and patients with concomitant injuries that needed further operative procedure under general anesthesia or spinal anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Intra-operative pain score | duration of operation
  pain assessment during operation at the following moments: before the injection, during injections , during the incision , during gentle manipulation , during aggressive manipulation and during wound closure.

SECONDARY OUTCOMES:
anaesthesia induction time | duration of operation
  the time taken to provide anesthesia
Blood loss | duration of operation
  calculated based upon the number and degree of soaking of swabs used in the operation and the amount in a suction container in the operation room.
intra-operative preserved motor power intraoperative | duration of operation
  surgeon test the motor power after repair of the affected tendon
operative time | duration of operation
  time from skin incision till last suture applied for wound closure
patient satisfaction | 12 hours post operative
  was measured and recorded using five-point Likert scale[25] (1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, and 5 = very satisfied) with checklist and a closed-ended question "If you were to undergo this surgery again, would you choose the same type of anaesthesia? YES or NO "
postoperative pain scores | 12 hours postoperatively
  numeric pain rating scale (NRS)A respondent selected a whole number (0- 10 integers) that best reflects the intensity of his pain, 0-10 was recorded by a blinded investigator at 2, 4, 6, 8, 10, 12 hours postoperatively, time of 1st call for postoperative analgesia was recorded, patients received 25 mg pethidine IV if the NRS pain exceeds 3, the dose was repeated on patient's demand with 2 hours minimal time interval between doses, total analgesic dose required in the 1st twelve hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Salwa O. Mohammed, M.D., Principal Investigator — Assistant professor, Ain Shams University, Faculty of Medicine
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No